CLINICAL TRIAL: NCT04938726
Title: Ketone Monoester Supplementation in Cystic Fibrosis: A Pilot and Feasibility Study
Brief Title: Ketone Supplementation in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eric P. Plaisance, Associate Professor and Chair, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300007323; P30DK079626 (NIH)
Record Dates: First submitted 2021-06-09; First posted 2021-06-24 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Two-way ANOVA with repeated measures on time
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All involved with blinded, except for the study pharmacist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone Monoester (Experimental): The ketone used is from KetoneAid and is commercially available as KE4 and will be consumed at 30 mL twice daily (15 g / dose)
  Interventions: Dietary Supplement: Ketone Monoester
- Placebo (Placebo Comparator): A placebo is being manufactured by KetoneAid to match the taste and other characteristics of the ketone supplement for blinding purposes
  Interventions: Dietary Supplement: Ketone Monoester

INTERVENTIONS:
Dietary Supplement: Ketone Monoester — Ketone supplement will be taken by mouth at a dose of 15 mL twice per day

SUMMARY:
This study will examine the effects of a novel ketone monester supplement on patients with cystic fibrosis experiencing an acute pulmonary exacerbation requiring hospitalization. Patients will undergo standard testing along with blood sampling to examine concentrations of inflammatory markers. Patients will then receive the ketone supplement for 5 days followed by post-testing to examine changes in pulmonary function and inflammatory markers

DETAILED DESCRIPTION:
Up to 25 hospitalized patients with cystic fibrosis will take part in this study at UAB. Patients will be randomly assigned to receive either an exogenous ketone or placebo supplement. Participants will take the ketone or placebo for 5 days during hospitalization. Participants will drink one 60 mL bottle twice daily of either the ketone or placebo. On day 1 and day 5, before the patient drinks the ketone (or placebo) the patient will be asked to fast overnight for 8 hours. Following administration of the first morning dose of ketones (or placebo) blood samples will be obtained from a finger stick before (time 0 min) and following (15, 30, 60, 90, and 120 min) after they drink the supplement. A commercially available ketone meter (Keto-Mojo, Napa, CA) that provides instant assessment of circulating ketone concentrations will be used to measure ketone concentrations in the blood. Medical history history will be obtained at hospitalization. The study team will also examine the body for any abnormal signs and symptoms. Sputum and blood will be collected prior to and following the ketone supplement or placebo. The hypothesis is that ketone supplementation will reduce inflammation via a well known inflammatory pathway to improve outcomes in patients with cystic fibrosis experiencing an acute pulmonary exacerbation

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF
* Age >19
* Colonization with P. Aeruginosa
* Acute pulmonary exacerbation requiring inpatient care

Exclusion Criteria:

* Concurrent or recent (within 28 d of enrollment) use of corticosteroids
* Inability to produce sputum
* Acute respiratory failure
* Chronic liver or renal disease
* Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Plaisance, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketone Monoester | Placebo
Started | 10 | 5
Completed | 9 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketone Monoester | Placebo | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 4 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Function Testing
Description: FEV1.0 (L/sec)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 9 | 5
L/sec | 1.9 (0.9) | 2.0 (1.0)

2. Primary Outcome: Inflammatory Markers
Description: Interleukin 1Beta (pg/mL)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 9 | 5
pg/mL | 0.3 (0.1) | 0.1 (0.1)

3. Secondary Outcome: Subjective Respiratory Quality of Life
Description: The Cystic Fibrosis Questionnaire-Revised (CFQ-R) was used to examine multiple domains related to quality of life. An outcome of the study was to examine subjective ratings of respiratory function using the CFQ-R comparing the ketone treated (KME) vs. control (placebo-control) groups.
  The measurement range for the score is from 0 - 100 with higher values representing a better outcome.
Time Frame: 5-7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 9 | 5
units on a scale | 70.1 (28.5) | 60.3 (26)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Ketone Monoester | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

LIMITATIONS AND CAVEATS:
Recruitment was difficult in this population because with the advent of CFTR modulators, patients are remarkably improved in health and have less incentive to participate in clinical studies outside of this domain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT04938726/Prot_000.pdf